CLINICAL TRIAL: NCT00156156
Title: A Phase 3, Continuation Study to Evaluate the Long-Term Safety of Asoprisnil in Subjects With Uterine Leiomyomata
Brief Title: Study of Asoprisnil in the Treatment of Uterine Fibroids.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-FB04-078
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Fibroid Uterus; Leiomyoma; Menorrhagia; Metrorrhagia; Uterine Fibroids
Keywords: Symptomatic Uterine Fibroids; Excessive Uterine Bleeding; Uterine Hemorrhage
MeSH Terms: conditions — Leiomyoma; Menorrhagia; Metrorrhagia; Uterine Hemorrhage | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil

INTERVENTIONS:
Drug: Asoprisnil — Asoprisnil 10 mg Tablet, oral Daily for up to 2 years
  Other Names: J867
  Arms: 1
Drug: Asoprisnil — Asoprisnil 25 mg Tablet, oral Daily for up to 2 years
  Other Names: J867
  Arms: 2

SUMMARY:
The objective of this study is to determine the long-term safety of asoprisnil in women with abnormal uterine bleeding associated with uterine fibroids.

DETAILED DESCRIPTION:
No medical therapy is currently available for the long-term treatment of abnormal uterine bleeding associated with uterine fibroids in women and many women must resort to surgery for relief. The objective of this study is to determine the long-term safety of two asoprisnil doses (10 and 25 mg tablets) administered daily to women who received asoprisnil in one of the asoprisnil long-term studies (study C03-062 or study M01-391). The safety endpoints for this study will include the affects of asoprisnil on the endometrium, ovaries, bone (a subset of study M01-391 subjects), lipid profiles, adverse events, and changes from baseline lab values and vital signs.

Some subjects receiving asoprisnil developed endometrial changes. As a result, dosing was prematurely discontinued for all subjects. To ensure safety, subjects will remain on study and will undergo scheduled study procedures. In most subjects, endometrial changes reversed after asoprisnil discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Women who have completed 12 months of active treatment in study M01-391 and Month 12 visit procedures Or completed 18 months of active treatment in study C03-062 and Month 18 visit procedures (with no more than a 14-day interruption in dosing from study C02-062 and this study) OR could not continue in a previous asoprisnil study, but are now eligible for retreatment
* Otherwise in good health
* Premenopausal based on Estrogen and FSH levels
* Adequate endometrial biopsy with no significant histological disorder
* Agrees to use double-barrier method of contraception

Exclusion Criteria:

* Any abnormal lab or procedure result(s) the study-doctor considers important
* History of a blood-clotting disorder
* History of osteoporosis requiring treatment
* Any invasive procedure(s) (D&C, etc) where a polyp was confirmed or a surgical or invasive procedure for uterine fibroids was performed during any previous asoprisnil study
* Hemoglobin < 8.0 g/dL
* Endometrial thickness ≥ 19 mm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2004-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Long-term Safety. | Throughout 2 year treatment period

SECONDARY OUTCOMES:
Change from baseline in the monthly bleeding score and the number of days with bleeding. | Each Month
Change from baseline in hemoglobin, hematocrit, TIBC, ferritin and iron concentrations. | Months 3, 6, 9,12,15,18, 24
Percent change from baseline in volume of the largest fibroid. | Months 12, 24
Change from baseline in bloating, pelvic pressure, dysmenorrhea and urinary symptoms. | Months 6, 12, 18, 24
Change from baseline in total symptom severity score and the Uterine Fibroid Symptoms-Quality of Life total score. | Months 6, 12, 18, 24
Change from baseline in the 8 scales of the SF-36 questionnaire. | Months 6, 12, 18, 24
Change from baseline in the 4 scales and overall index of the Work Limitations Questionnaire. | Months 6, 12, 18, 24
Cumulative percent of subjects who achieve amenorrhea. | Each Month

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott